CLINICAL TRIAL: NCT04437719
Title: Longitudinal Prospective Cohort Study to Describe the Clinical Characteristics of COVID-19, the Acquired Immune Response and the Biological and Clinical Parameters of Patients Followed in Oncology by the Saint-Joseph Hospital Group, Paris, France for a Period of 6 Months During the COVID-19 Pandemic in 2020
Brief Title: Prospective Cohort Study to Describe the Clinical Characteristics of COVID-19, the Acquired Immune Response and the Biological and Clinical Parameters of Patients Followed in Oncology by the Saint-Joseph Hospital Group for a Period of 6 Months During the COVID-19 Pandemic
Acronym: OBVIONCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: ObvioHealth (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OBVIONCO
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Oncology; COVID-19
MeSH Terms: conditions — Neoplasms; COVID-19

STUDY DESIGN:
Intervention Model Description: As part of this research, the patient must complete questionnaires daily on the Obvio-19 application, one of 5 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obvio-19 App (Experimental): If the patient is willing to participate to the trial, his given oral, free, informed and express consent will be collected and traced in his medical file. After enrollment, patients will be sent an invitation via email to download the Obvio-19 mobile app. After downloading the Obvio-19 app, patients will receive instructions as to how they may communicate with the study investigator. Communication may occur through the chat function of the app or live telephone conversations.
  Patients must log into the Obvio-19 app daily to complete the questionnaires. The Obvio-19 system is designed to identify responses that indicate the participant is at an increased risk for serious illness or exhibiting serious symptoms, such as coughing up blood. Such patients will be notified by the app of this status and prompted to seek medical attention.
  Interventions: Other: Obvio-19 app

INTERVENTIONS:
Other: Obvio-19 app — As part of this research, the patient must complete questionnaires daily on the Obvio-19 application, one of 5 minutes.
  Evaluation of the proportion of patients with COVID-19 infection's symptoms known to be associated with COVID-19 diagnosis (fever, cough, loss of taste and smell, sore throat, muscle pain, diarrhea, fatigue, difficulty eating and drinking and shortness of breath) followed during a period of 6 months.
  To assess the prevalence and course of symptoms of COVID-19 infection of patients followed during a period of 6 months.
  To establish the correlation of the COVID-19 infection with the biological and clinical data of patients from the Oncology cohort of the Groupe hospitalier Paris Saint-Joseph in Paris followed during a period of 6 months.

SUMMARY:
This registry will allow to evaluate the correlation of the incidence and evolution of associated symptoms of infection of COVID-19 with the biological and clinical parameters in patients followed in Oncology during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Prior to conducting any of the screening tests, the Investigator or his designee will explain the trial fully to the prospective patient and provide him with a copy of the Patient Information Leaflet/Informed Consent Form.

If the patient is willing to participate to the trial, his given oral, free, informed and express consent will be collected and traced in his medical file.

The screening questionnaire will be completed. The patient's suitability for the trial will be confirmed by the inclusion/exclusion criteria .

Following completion of the Baseline Questionnaire, patients will receive the Daily Questionnaire. This is designed to assess if they have developed symptoms associated with COVID-19 infection.

If a participant responds that they are not feeling well, a series of follow-up questions will be asked regarding what symptoms they are currently experiencing.

The Daily Questionnaire will be asked of patients every day throughout the Observation Period of 6 months.

At the end of the Observation Period, all patients will complete a series of questionnaires relating to the conduct of the study and tools employed.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient followed in the medical oncology department of Paris Saint-Joseph Hospital Paris in France
* Patient Having regular access to smartphone and internet sufficient to support study demands
* French-speaking patient
* Affiliation to the social security network
* Willing and able to provide given oral, free, informed and express consent

Exclusion Criteria:

* Patients unable or unwilling to perform all requested study tasks
* Patient under tutorship or curatorship
* Patient deprived of liberty
* Pregnant or lactating patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
COVID-19 infection's symptoms | Observational period of 6 months
  Evaluation of the proportion of patients with COVID-19 infection's symptoms known to be associated with COVID-19 diagnosis (fever, cough, loss of taste and smell, sore throat, muscle pain, diarrhea, fatigue, difficulty eating and drinking and shortness of breath) followed during a period of 6 months.

SECONDARY OUTCOMES:
Incidence and course of symptoms of COVID-19 infection | During a period of 6 months
  To assess the prevalence and course of symptoms of COVID-19 infection of patients followed during a period of 6 months.
Correlation of the COVID-19 infection with the biological and clinical data of patients | After a period of 6 months
  To establish the correlation of the COVID-19 infection with the biological and clinical data of patients from the Oncology cohort of the Groupe hospitalier Paris Saint-Joseph in Paris followed during a period of 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Raymond, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Result] Gliklich RE, Dreyer NA, Leavy MB, Christian JB, editors. 21st Century Patient Registries: Registries for Evaluating Patient Outcomes: A User's Guide: 3rd Edition, Addendum [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2018 Mar. Report No.: 17(18)-EHC013-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK493818/ PMID 29708678
- See also: Features, Evaluation and Treatment Coronavirus (COVID-19) Marco Cascella; Michael Rajnik; Arturo Cuomo; Scott C. Dulebohn; Raffaela Di Napoli. — https://www.ncbi.nlm.nih.gov/books/NBK554776/